CLINICAL TRIAL: NCT01334359
Title: ERPs to Academics: Exercise Effects on Cognition in School-Aged Children
Brief Title: Exercise Effects on Cognition in School-Aged Children
Acronym: FITKids
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Principal Investigator, Chuck Hillman, Professor, University of Illinois at Urbana-Champaign
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 1R01HD055352-01A2 (NIH)
Record Dates: First submitted 2011-04-08; First posted 2011-04-13 (Estimated); Last update posted 2014-07-25 (Estimated); Status verified 2014-07

CONDITIONS: Brain Health; Cognition; Scholastic Achievement
Keywords: physical activity; fitness; brain health; cognition; scholastic achievement; preadolescent children
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment Group (Experimental): Participants randomized to the afterschool intervention
  Interventions: Behavioral: Physical Activity
- Wait List Group (Placebo Comparator): Participants in this group partake in their regular afterschool activities, without intervention from the study staff.
  Interventions: Behavioral: Physical Activity

INTERVENTIONS:
Behavioral: Physical Activity — 9-month afterschool program designed to increase physical activity and aerobic fitness.

SUMMARY:
Recent trends have identified decreasing levels of physical activity, fitness, and health in preadolescent children. Examining factors, such as physical activity behavior and aerobic fitness that positively influence cognitive health of school-age children are important for improving school performance, maximizing health, and improving the overall functioning of individuals as they progress through the human lifespan. A sample of preadolescent children from the Urbana, Illinois elementary school system will be randomly assigned to a 9- month afterschool program that focuses on either aerobic exercise or wait-list control group to determine the effects of physical activity on basic and applied aspects of cognition. Changes in neuroimaging and behavioral indices of cognitive function and performance on standardized academic achievement tests of mathematics and reading will be examined as a function of participation in the intervention. Preliminary research supports that physical activity is positively associated with basic and applied aspects of cognition, with a stronger relationship for tasks requiring extensive amounts of executive control. However, previous research has mainly focused on older adults, and little research has examined the relationship between physical activity and executive control in children. These findings will provide lifestyle considerations for children to improve their cognitive health across the lifespan.

DETAILED DESCRIPTION:
The aim of this proposal is to improve our understanding of factors related to brain health and cognition of school-aged children by examining the effects of a 9-month exercise intervention on basic and applied aspects of cognition in preadolescent children. From a basic measurement perspective, event-related brain potentials, MRI, fMRI, and behavioral indices of cognition will be studied during several tasks aimed at assessing various aspects of executive control. Preliminary research has observed faster and more efficient performance in high-fit, relative to low-fit, children and adults using neuroelectric measures that reflect attentional allocation to environmental stimuli and response monitoring processes, along with behavioral measures that reflect response speed and accuracy. These preliminary findings indicate greater top-down attentional control may be associated with increases in physical activity. From an applied measurement perspective, preliminary research has found that children with greater aerobic fitness perform better on standardized achievement tests of reading and mathematics, compared to children with lower aerobic fitness, suggesting that exercise may be related to academic performance in an applied school setting. To date, no causal evidence exists regarding the effects of physical activity on neuroelectric, behavioral, or applied school performance indices of cognition in children. Accordingly, this proposal investigates an aerobic activity training intervention on these measures of cognition using three tasks that require variable amounts of executive control, and on the Illinois Standardized Achievement Test using a randomized control design in which participants are assigned to an afterschool physical activity program or a wait-list control group. Given recent trends identifying decreased levels of physical activity and health status in preadolescents, the understanding of the potential benefits of physical activity on cognition is of great interest. It is imperative that factors positively influencing cognitive function of children be examined to maximize health and effective functioning of individuals as they progress through the lifespan.

ELIGIBILITY:
Inclusion Criteria:

* Parental consent
* 7.5-9.5 years
* Capable of performing exercise
* Absence of school-identified learning disability
* IQ > 85
* Tanner Scales score <= 2
* ADHD Rating Scales score > 85%

Exclusion Criteria:

* Non-consent of guardian
* Above or Below age range
* Any physical disability that prohibits exercise
* School-identified learning disability
* IQ < 85
* Tanner Scales Score > 2
* ADHD Rating Scale score < 85%

Ages: 8 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 252 (Actual)
Dates: Start 2008-07; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Event-related brain potentials | Change from baseline, 36-40 weeks
  Measures of the neuroelectric system that occur in response to, or in preparation for, a discrete event.
Task Performance | Change from baseline, 36-40 weeks
  Measures of responses speed and accuracy
Academic Achievement | Change from baseline, 36-40 weeks
  Scholastic achievement tests of reading comprehension and arithmetic.

SECONDARY OUTCOMES:
Magnetic Resonance Imaging | Change from baseline, 36-40 weeks
  Measures of brain structure.
functional Magnetic Resonance Imaging | Change from baseline, 36-40 weeks
  measures of brain function
Eye Tracking | Change from baseline, 36-40 weeks
  Measures of visual gaze.
Virtual Reality | Change from baseline, 36-40 weeks)
  Measures of response speed and accuracy related to crosswalk behavior
Adiposity | Change from baseline, 36-40 weeks
  Measure of change in adiposity
Diet and Brain Function | Change from baseline, 36-40 weeks
  Measure of correlation between diet and brain function

CONTACTS AND LOCATIONS:
Overall Officials: Charles H Hillman, PHD, Principal Investigator — University of Illinois at Urbana-Champaign
Locations (1):
- University of Illinois, Urbana, Illinois, United States

REFERENCES:
- [Derived] Logan NE, Westfall DR, Raine LB, Anteraper SA, Chaddock-Heyman L, Whitfield-Gabrieli S, Kramer AF, Hillman CH. The Differential Effects of Adiposity and Fitness on Functional Connectivity in Preadolescent Children. Med Sci Sports Exerc. 2022 Oct 1;54(10):1702-1713. doi: 10.1249/MSS.0000000000002964. Epub 2022 Jun 24. PMID 35763600
- [Derived] Chojnacki MR, Holscher HD, Balbinot AR, Raine LB, Biggan JR, Walk AM, Kramer AF, Cohen NJ, Hillman CH, Khan NA. Relations between mode of birth delivery and timing of developmental milestones and adiposity in preadolescence: A retrospective study. Early Hum Dev. 2019 Feb;129:52-59. doi: 10.1016/j.earlhumdev.2018.12.021. Epub 2019 Jan 12. PMID 30641478
- [Derived] Raine LB, Khan NA, Drollette ES, Pontifex MB, Kramer AF, Hillman CH. Obesity, Visceral Adipose Tissue, and Cognitive Function in Childhood. J Pediatr. 2017 Aug;187:134-140.e3. doi: 10.1016/j.jpeds.2017.05.023. Epub 2017 Jun 13. PMID 28622956
- [Derived] Hillman CH, Pontifex MB, Castelli DM, Khan NA, Raine LB, Scudder MR, Drollette ES, Moore RD, Wu CT, Kamijo K. Effects of the FITKids randomized controlled trial on executive control and brain function. Pediatrics. 2014 Oct;134(4):e1063-71. doi: 10.1542/peds.2013-3219. PMID 25266425
- [Derived] Khan NA, Raine LB, Drollette ES, Scudder MR, Pontifex MB, Castelli DM, Donovan SM, Evans EM, Hillman CH. Impact of the FITKids physical activity intervention on adiposity in prepubertal children. Pediatrics. 2014 Apr;133(4):e875-83. doi: 10.1542/peds.2013-2246. Epub 2014 Mar 31. PMID 24685956
- [Derived] Baym CL, Khan NA, Monti JM, Raine LB, Drollette ES, Moore RD, Scudder MR, Kramer AF, Hillman CH, Cohen NJ. Dietary lipids are differentially associated with hippocampal-dependent relational memory in prepubescent children. Am J Clin Nutr. 2014 May;99(5):1026-32. doi: 10.3945/ajcn.113.079624. Epub 2014 Feb 12. PMID 24522447